CLINICAL TRIAL: NCT01950832
Title: Evaluation of the Macula, Retinal Nerve Fiber Layer and Choroid Thickness in Women With Polycystic Ovary Syndrome By Using Spectral-domain Optical Coherence Tomography.
Brief Title: Eye Evaluation in Patients With PCOS
Status: Completed | Type: Observational
Sponsor: Gökhan Açmaz (Other Government)
Responsible Party: Sponsor-Investigator, Gökhan Açmaz, MD, Kayseri Education and Research Hospital
Organization: Kayseri Education and Research Hospital (Other Government)
Other Study IDs: Gökhan Açmaz; Kayseri ERH (Other: Kayseri Education and Research Hospital)
Record Dates: First submitted 2013-09-17; First posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: PCOS
Keywords: Structure of Retina; Macular Thickness; Retinal Nerve Fiber Layer; Choroidal Thickness; PCOS; Optical Coherence Tomography
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- polycystic ovary syndrome (PCOS) group: Patients who were diagnosed as PCOS according to 2003 Rotterdam Criteria.
  Interventions: Other: Investigating clinically normal patients with optic coherence tomography
- Control: 60 healthy volunteers
  Interventions: Other: Investigating clinically normal patients with optic coherence tomography

INTERVENTIONS:
Other: Investigating clinically normal patients with optic coherence tomography
  Other Names: Control Group

SUMMARY:
To evaluate the macular, retinal nerve fiber layer (RNFL) and choroidal thickness alterations by using spectral-domain optical coherence tomography (SD-OCT) in polycystic ovary syndrome (PCOS) and to compare them with healthy reproductive-age women controls.

DETAILED DESCRIPTION:
PCOS was diagnosed according to Rotterdam criteria that include (i) oligomenorrhea (interval between periods was ≥35 days) or amenorrhea (absence of vaginal bleeding for 6 months); (ii) hyperandrogenism; (iii) polycystic ovaries and exclusion of other PCOS-like syndromes, such as adrenal dysfunction, Cushing's syndrome, congenital adrenal hyperplasia, androgen-secreting tumors, enzyme deficiency (21-hydroxylase in particular), hyperprolactinemia, and thyroid dysfunction. Ultrasonographic diagnosis of polycystic ovaries was based on the presence of multiple cysts (≥12 small follicles in each ovary [2-9 mm in diameter]) arranged peripherally and scattered throughout the dense core of stroma (the necklace appearance of follicular cysts), and/or increased ovarian volume >10 ml on pelvic or vaginal ultrasound examination.

Patients who were allocated in control group had regular menstrual cycle and normal ovarian morphology detected by ultrasounds. None of the participants in both groups were pregnant. All patients were evaluated in follicular phase of their menstrual cycle.

Each subject underwent a comprehensive ophthalmologic examination. Following this detailed ophthalmologic examination, the third-generation Spectralis OCT device was used for the assessment. The OCT assessments of involved in the study were performed by the same experienced technician. The procedure was achieved without pupillary dilatation and under the same intensity of dim room lighting.

Macular thickness was determined automatically and was analyzed by OCT software. Fast Macular Thickness Map option was utilized for the macular measurements. During the assessments, macular thickness and volume analysis were used. We selected the macular map analysis protocol on the Spectralis to display numeric averages of the measurements for each of the 9 subfields as defined by the Early Treatment Diabetic Retinopathy Study (ETDRS) The peripapillary RNFL thickness parameters that were automatically calculated by the fast RNFL mode and divided into regions included temporal quadrant thickness, temporal superior quadrant thickness, nasal superior quadrant thickness, nasal quadrant thickness, nasal inferior quadrant thickness, temporal inferior quadrant thickness, and average thickness.

The method of obtaining enhanced depth imaging (EDI) OCT images has been reported previously. The resultant images were viewed and measured with the contained Heidelberg Eye Explorer software. Choroid imaging was obtained by activating the EDI button. The choroid was manually measured from the outer border of the hyperreflective line corresponding to the retinal pigment epithelium to the inner surface of the sclera. The measurements of subfoveal choroidal thickness were done by one of the authors in a masked fashion without knowledge of subject information.

ELIGIBILITY:
Inclusion Criteria:

Patients who were diagnosed as PCOS according to 2003 Rotterdam Criteria, had no physical disease but PCOS, did not receive any treatment for 6 months prior to the study for PCOS or for co-morbidities and had at least primary school degree.

Exclusion Criteria:

Patients who had thyroid disorders, hypertension, thromboembolic disease, diabetes mellitus, cardiovascular events, Cushing' disease, positive malignancy, congenital adrenal hyperplasia, liver disease,psychotic disorders and used antidepressants or steroidal hormone drugs and mood stabilizers (Li, Valproic acid, COCs, antiandrogens or insulin sensitizers etc.)

Ages: 16 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants:
  Patients who were diagnosed with PCOS according to 2003 Rotterdam Criteria, had no physical disease but PCOS, did not receive any treatment for 6 months prior to the study for PCOS or co-morbidities and had at least primary school degre will enroll into the study. The second group consisted of 60 healthy volunteer participants in reproductive age.
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Macula, Retinal nerve fiber and choroid layer measurements | 1 month
  Each subject underwent a comprehensive ophthalmologic examination. Following this detailed ophthalmologic examination, the third-generation Spectralis OCT device (software version 5.6.3.0; Spectralis OCT Heidelberg Engineering, Dossenheim, Germany) was used for the assessment. The OCT assessments of involved in the study were performed by the same experienced technician. The procedure was achieved without pupillary dilatation and under the same intensity of dim room lighting.

SECONDARY OUTCOMES:
Macular thickness and volume | 1 month
  Central subfield, inferior inner macula, inferior outer macula, nasal inner macula, nasal outer macula, superior inner macula, superior outer macula, temporal inner macula, temporal outer maculas both thickness and volumes were evaluated.

OTHER OUTCOMES:
Retinal nerve fiber layer and choroid measurements. | 1 month
  Temporal Superior, nasal Superior, nasal, nasal Inferior, temporal inferior parts of RNFL were evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Açmaz, MD, Principal Investigator — Kayseri Education and Research Hospital
Locations (1):
- Kayseri Education and Research Hospital, Kayseri, Turkey (Türkiye)